CLINICAL TRIAL: NCT03813654
Title: Sleep and Circadian Treatments for Shift Workers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for project ended
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Massachusetts, Lowell (Other)
Responsible Party: Principal Investigator, Jeanne Duffy, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-P-002341; R01AG044416 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-23 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Shift-Work Sleep Disorder; Shift-Work Related Sleep Disturbance
Keywords: sleep; attention; vigilance; aging; shift work
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: The interventional study design describes the Field Trial only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Group A) (No Intervention): During the intervention block of the Field Trial, at the end of the first night shift, the participant will be told about their randomization group. In the control group (Group A), participants will not be given any instructions about the timing or duration of their sleep, but will be instructed to follow their usual night shift sleep routine.
- 8-h Afternoon-Evening Sleep (Group B) (Experimental): In the 8-h afternoon-evening sleep intervention group (Group B), participants will be instructed to go to bed between 13:00 and 14:00 (depending on their individual commute time) and to remain in bed attempting to sleep for 8 hours (until 21:00-22:00) before the next two night shifts.
  Interventions: Behavioral: 8-h Afternoon-Evening Sleep
- 8-h Free Sleep (Group C) (Experimental): In the 8-h free sleep group (Group C), participants will be instructed to remain in bed for 8 continuous hours before the next two night shifts, but will not be given any instruction regarding which 8 hours they should sleep.
  Interventions: Behavioral: 8-h Free Sleep

INTERVENTIONS:
Behavioral: 8-h Afternoon-Evening Sleep — 8 consecutive hours time in bed during the afternoon/evening.
  Arms: 8-h Afternoon-Evening Sleep (Group B)
Behavioral: 8-h Free Sleep — 8 consecutive hours time in bed at any time.
  Arms: 8-h Free Sleep (Group C)

SUMMARY:
There are three components to this study: a Field Trial, a Shift Worker Survey, and Focus Groups. The Investigators will study the effectiveness, feasibility, and acceptability of an 8-h sleep intervention in older night workers in an operational environment. The overall goal of the Field Trial is to minimize sleep deficiency and negative outcomes resulting from that, including sleepiness and performance impairments during night shift work. The Shift Worker Survey is designed to understand some of the demographic and operational factors that enable or inhibit the ability of individual shift workers to adopt this intervention. The Focus Groups are designed to glean in-depth information from older shift workers who indicate that they are unable or unwilling to adopt an 8-h sleep timing intervention. Understanding these factors will assist in refining and targeting the intervention to those individuals who will be most likely to benefit from the intervention sleep timing strategy.

DETAILED DESCRIPTION:
The overall goal of the Field Trial is to minimize sleep deficiency and negative outcomes resulting from that, including sleepiness and performance impairments during night shift work. The experimental protocol is divided into two blocks, the Baseline block and the Intervention block, where participants will work at least 3 night shifts in a row within each block. For at least one week prior to the baseline block participants will work their usual shift schedule (i.e., no vacation/scheduled days off). The investigators will recruit up to 200 health care workers in order to have up to 75 health care workers complete the entire Field Trial. Potential participants will be employed older health care workers who work a minimum number of 8-h night shifts per month and who are in the greater Boston area.

The Shift Worker Survey is designed to understand some of the demographic and operational factors that enable or inhibit the ability of individual shift workers to adopt the sleep intervention that will be tested in the Field Trial. The investigators will use a web-based survey consisting of ~70 questions developed and administered using REDCap. The complete questionnaire will take approximately 20-30 minutes to complete. The study will enroll up to 1,000 employed individuals (20 or more hours per week) whose work includes overnight shifts, with a minimum criterion of at least 4 night shifts a month. Health Care Workers who complete the Shift Worker Survey will be given the option to complete an additional Health Care Worker's Questionnaire at the end of the basic Shift Worker Survey. Those whose responses meet inclusion/exclusion criteria for the Field Trial will be informed at the end of the Shift Worker Survey that they may be eligible for the Field Trial.

The goal of the Focus Groups is to gain information on the feasibility and acceptability of the fixed 8-h sleep schedule from the participants' perspective. Investigators will seek to learn more information about the current sleep strategies they use on a regular basis, and both the facilitating and challenging aspects of the fixed-sleep countermeasure (e.g., individual, intrapersonal and organizational barriers to implementation of fixed 8-h sleep, recommended modifications to the fixed 8-h sleep schedule that would make it more user-friendly while maintaining scientific validity). Each of the focus groups will consist of 4-6 individuals to stimulate discussion without leaving participants out, and will last 60-90 minutes. The investigators aim to enroll up to 60 individuals in Focus Groups. In addition to the health care workers who took part in the Field Trial, the investigators will invite night shift workers who complete the Shift Worker Survey but indicate their inability to comply with a fixed 8-h sleep schedule to attend a Focus Group discussion.

ELIGIBILITY:
Field Trial -

Inclusion Criteria:

* Age 50-65 years
* Health care workers who work a minimum of 4 night shifts (8-4) per month
* Must live in the greater Boston area
* Must report an ability to work three successive 8-h night shifts during two weeks
* Must report an ability to spend 8 consecutive hours in bed attempting to sleep prior to the final two successive night shifts in the second study week
* Must have a typical commute time between home and place of work of less than one hour

Exclusion Criteria:

* Non-optional activities that would interfere with the participant's ability to remain in bed attempting to sleep if randomized to an 8-h sleep group
* Prescription or over-the-counter medication(s) known to affect sleep [e.g., hypnotics] or alertness [e.g., antihistamines]

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne F Duffy, MBA, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between September 2019 and November 2022. All recruitment was via advertisements placed online, in newsletters, and through email lists.
Pre-assignment Details: Enrollment was assigned upon start of the Baseline period, but participants were not informed of their randomization until after the first night shift of the Intervention period.
Period: Overall Study
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Started | 11 | 11 | 11
Completed | 10 | 10 | 9
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C) | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 9 | 29
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (4.2) | 58.3 (5) | 58.6 (2.9) | 56.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 7 | 23
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 9 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 9 | 8 | 8 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 29
Years Working Night Shifts [Number; unit: participants] — Years by participant report.
  participants
    less than 1 year | 1 | 0 | 1 | 2
    1-5 years | 1 | 1 | 1 | 3
    6-10 years | 1 | 1 | 1 | 3
    11-24 years | 3 | 5 | 2 | 10
    more than 25 years | 4 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (TST)
Description: TST is calculated as minutes of sleep in the main sleep episode between shifts, derived from actigraphy data collected in 60 s epochs. The investigators will use a commercial software package to score the sleep. For control group participants who will sleep ad-lib, TST will be calculated for the major sleep episode but also will be summed across sleep episodes if they sleep in more than one bout.
Time Frame: The TST averaged for up to 3 intervention nights (in minutes) will be compared between groups.
Population: All participants with useable actigraphy data were included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 8
minutes | 338 (68.7) | 387 (53.2) | 428 (66.7)
Statistical Analysis 1: Comparison: Control (Group A) vs 8-h Afternoon-Evening Sleep (Group B) vs 8-h Free Sleep (Group C); Test type: Other — Mixed model analysis with post-hoc tests; p < 0.05, Mixed Models Analysis — A priori threshold was <0.05; Mean Difference (Final Values) = 90, Standard Deviation 68.7 — This is the difference between the control and 8-h Free Sleep Group

2. Primary Outcome: Sleep Fragmentation Index (FI)
Description: FI will be calculated as the number of times that sleep was terminated after 1 minute, expressed as a percentage of total estimated sleep time, using actigraphy data and commercial software to calculate it.
Time Frame: The FI averaged for intervention nights 2 and 3 will be compared between groups.
Population: All participants with useable actigraphy data were included.
Measure: Mean (Standard Deviation); unit: percentage of TST
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 7
percentage of TST | 22.15 (15.49) | 34.94 (22.01) | 29.25 (15.45)

3. Primary Outcome: Wake After Sleep Onset (WASO)
Description: WASO is an objective sleep quality measure and will be calculated as the duration (in minutes) of all awakenings during the main sleep episode measured with actigraphy, and calculated using commercial software.
Time Frame: The WASO averaged for intervention nights 2 and 3 will be compared between groups.
Population: All participants with useable actigraphy data were included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 7
minutes | 38.85 (32.69) | 83.18 (57.96) | 70.06 (43.6)

4. Primary Outcome: Subjective Sleep Quality
Description: Participants will report their subjective sleep quality daily upon awakening from the main sleep episode. Multiple measures of subjective sleep quality will be assessed, but the investigators will report how refreshed the participant feels after awakening as the outcome. This is rated on a 7-point scale, where 7 is the best and 1 is the worst.
Time Frame: Subjective Sleep quality (refreshment) averaged for intervention nights 2 and 3 will be compared between groups.
Population: Every participant with responses at waketime after night shifts 2 and/or 3 during the intervention segment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 8
units on a scale | 3.25 (1.03) | 3.06 (1.36) | 3.13 (0.88)

5. Primary Outcome: Subjective Alertness Via Karolinska Sleepiness Scale (KSS)
Description: Participants will complete the Karolinska Sleepiness Scale (KSS) as a measure of subjective alertness immediately following each night shift. The KSS is a Likert scale ranging from 1, extremely alert, to 9, extremely sleepy.
Time Frame: The KSS score taken at the end of the final night shift (night shift 3) during the intervention block will be compared to that at baseline.
Population: All participants completing the study for whom data were available.
Measure: Number; unit: participants
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 9 | 7 | 9
participants
  subjective sleepiness worsened between baseline and end of treatment | 5 | 0 | 3
  subjective sleepiness did not change between baseline and end of treatment | 3 | 3 | 4
  subjective sleepiness improved between baseline and end of treatment | 1 | 4 | 2

6. Primary Outcome: Sustained Attention
Description: The psychomotor vigilance task (PVT) is a test of visual reaction time (RT) in which the participant is asked to maintain the fastest possible RTs to a simple visual stimulus for several minutes. The inter-stimulus interval varies randomly between 2-10 seconds. While there are a number of standard performance metrics that can be obtained from each PVT, we have looked at the slowest 10% of responses.
Time Frame: PVT mean of slowest 10% of responses measured at the start of the final night shift (night shift 3) during the intervention block will be compared between groups.
Population: There were many missing data for this outcome. Group A only had 1 participant in whom complete PVT results were available for the final night shift. Thus, no standard deviation is provided.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 1 | 10 | 5
milliseconds | 308.75 (0) | 393.27 (87.34) | 470.96 (126.80)
Statistical Analysis 1: Comparison: 8-h Afternoon-Evening Sleep (Group B) vs 8-h Free Sleep (Group C); We compared the PVT taken at the start of the final night shift between Group B and those in Group C who slept in the morning and had complete data. Our hypothesis was that Group B would have faster RTs; Test type: Superiority; p = 0.09, t-test, 1 sided — The groups had unequal variances, so we adjusted for unequal variances when doing the t-test. The a priori threshold for statistical significance was p<0.05; Adjusted for unequal variances between the two groups

7. Primary Outcome: Subjective Energy
Description: A Visual Analogue Scale (VAS) will be used to assess subjective energy level. The VAS consists of a 100mm horizontal line with each end of the line labeled with the extremes of a subjective continuum, e.g. energetic-sluggish. The Participant indicates a position on the line that best describes how they feel at that moment. Distance from the left end of the scale (0) to the indicated point will be measured in mm and reported as subjective energeticness. Thus, scores on the scale range from 0 to 100 with lower scores indicating greater subjective energy.
Time Frame: Subjective Energy measurements taken at the end of the final night shift (night shift 3) in the intervention block will be compared between groups.
Population: All participants who had data collected at the end of Intervention Night Shift 3.
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 9
units on a scale of 0-100 | 50.07 (27.17) | 57.72 (28.95) | 52.07 (22.53)

8. Primary Outcome: Subjective Stress Via Visual Analog Scale (VAS)
Description: A Visual Analogue Scale (VAS) will be used to assess subjective stress.The VAS consists of a 100mm horizontal line with each end of the line labeled with the extremes of a subjective continuum, e.g. relaxed-stressed. The Participant indicates a position on the line that best describes how they feel at that moment. Distance from the left end of the scale (0) to the indicated point will be measured in mm and reported as Subjective Stress. Thus, scores on the scale range from 0 to 100 with higher scores indicating greater subjective stress.
Time Frame: Subjective Stress via VAS measurements taken at the end of the final night shift (night shift 3) in the intervention block will be compared between groups.
Population: All participants who had data collected at the end of intervention night shift 3.
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 9
units on a scale of 0-100 | 58.99 (32.33) | 68.84 (20.29) | 76.52 (19.53)

9. Primary Outcome: Subjective Calmness Via Visual Analog Scale (VAS)
Description: A Visual Analogue Scale (VAS) will be used to assess subjective Calmness. The VAS consists of a 100mm horizontal line with each end of the line labeled with the extremes of a subjective continuum, e.g. calm-excited. The Participant indicates a position on the line that best describes how they feel at that moment. Distance from the left end of the scale (0) to the indicated point will be measured in mm and reported as Subjective Calmness. Thus, scores on the scale range from 0 to 100 with lower scores indicating greater subjective calmness.
Time Frame: Subjective Calmness via VAS measurements taken at the end of the final night shift (night shift 3) in the intervention block will be compared between groups.
Population: All participants who had data collected at the end of the 3rd Night Shift.
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 9
units on a scale of 0-100 | 80.14 (19.64) | 78.34 (15.42) | 78.51 (14.54)

10. Primary Outcome: Subjective Health Via Visual Analog Scale (VAS)
Description: Visual Analogue Scales (VAS) will be used to assess subjective health. VAS consist of a 100mm horizontal line with each end of the line labeled with the extremes of a subjective continuum, e.g. healthy-sick. The Participant indicates a position on the line that best describes how they feel at that moment. Distance from the left end of the scale (0) to the indicated point will be measured in mm and reported as Subjective Health. Thus, scores on the scale range from 0 to 100 with lower scores indicating greater subjective health.
Time Frame: Subjective Health via VAS measurements taken at the end of the final night shift (night shift 3) in the intervention block will be compared between groups.
Population: All participants who had data from the end of Intervention Night Shift 3.
Measure: Mean (Standard Deviation); unit: units on a scale of 0-100
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 10 | 9 | 9
units on a scale of 0-100 | 75.08 (15.12) | 78.88 (19.05) | 74.96 (16.78)

11. Primary Outcome: Subjective Alertness Via Visual Analog Scale (VAS) - DATA NOT COLLECTED
Description: Participants will complete the Visual Analog Scale (VAS) as a measure of subjective alertness three times per night shift: Once just before the night shift, once during their shift break, and once immediately following the night shift. The VAS consists of a 100mm horizontal line with each end of the line labeled with the extremes of a subjective continuum, e.g. sleepy-alert. Participants will indicate a position on the line that best describes how they feel at that moment. Distance from the left end of the scale to the indicated point will be measured in mm and reported as Subjective Alertness with higher scores indicating greater subjective alertness.
Time Frame: Subjective Alertness via VAS measurements taken at the end of the final night shift (night shift 3) in the intervention block will be compared between groups.
Population: These data are similar enough to measures from the Karolinska Sleepiness Scale data and in order to reduce participant burden WE DID NOT COLLECT THEM. We did not modify the IRB protocol to indicate this measure would not be collected. BECAUSE THEY WERE NOT COLLECTED WE CANNOT ANALYZE ANYTHING.
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Fatigue and Inter-Shift Recovery
Description: The Occupational Fatigue Exhaustion Recovery Scale (OFER 15), which consists of 15 questions about acute fatigue and recovery between shifts, will be used. Each of the 15 questions is answered on a Likert scale which ranges from 0 (Strongly Disagree) to 6 (Strongly Agree). The OFER15 will be completed immediately after the third night shift in the Baseline block and at the end of the third night shift in the Intervention block.
Time Frame: OFER15 scores from the end of the third night shift in the Baseline to the end of the Intervention block will be compared between groups.
Population: All participants who completed the study and who had complete questionnaire results from the Baseline and Intervention.
Measure: Number; unit: participants
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 8 | 6 | 8
participants
  Participants whose fatigue scores worsened between baseline and end of intervention. | 3 | 2 | 4
  Participants whose fatigue scores improved between baseline and end of intervention. | 5 | 4 | 4
  Participants whose refreshment scores worsened between baseline and end of intervention. | 3 | 3 | 7
  Participants whose refreshment scores did not change between baseline and end of intervention. | 0 | 1 | 0
  Participants whose refreshment scores improved between baseline and end of intervention. | 5 | 2 | 1

13. Secondary Outcome: Subjective Stress
Description: The investigators will collect subjective measures of daily stress using a validated questionnaire, the Perceived Stress Scale (PSS), a 10-item self-report measure that allows a person to indicate stressful events that they have experienced in the past week. Each question is answered on a 5-item scale indicating the frequency, from 1 (never) to 5 (very often).
Time Frame: Subjective stress will be assessed immediately after the third night shift in the Baseline and Intervention blocks and the change will be compared between groups.
Population: All participants who completed the study and who had Baseline and Intervention data.
Measure: Number; unit: participants
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 9 | 6 | 9
participants
  participants whose perceived stress worsened from baseline to end of intervention. | 3 | 3 | 2
  participants whose perceived stress did not change from baseline to end of intervention. | 1 | 1 | 2
  participants whose perceived stress improved from baseline to end of intervention. | 5 | 2 | 5

14. Secondary Outcome: Subjective Quality of Life: WHOQOLBref
Description: The investigators will use a validated questionnaire, the WHOQOLBref, a 26 item questionnaire suitable for field studies, which asks a series of questions about life, health, energy, and personal satisfaction, to assess Quality of Life. The questionnaire contains 4 separately scored domains: Physical Health, Psychological, Social Relationships, and Environment. Each domain contains several questions and ask participants to provide a response on a Likert Scale ranging from 1 to 5, with higher numbers indicating a higher quality of life (aside from 3 negatively phrased items).
Time Frame: WHOQOL-Bref will be taken at Baseline and immediately after the third night shift in the Intervention block and will be compared between groups.
Population: All participants who completed the study and who had baseline and end of intervention data.
Measure: Number; unit: participants
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 9 | 6 | 9
participants
  participants whose QOL score declined from baseline to end of intervention. | 5 | 2 | 3
  participants whose QOL score did not change from baseline to end of intervention. | 2 | 3 | 1
  participants whose QOL score improved from baseline to end of intervention. | 2 | 1 | 5

15. Secondary Outcome: Salivary Cortisol Level NOTE THAT THIS AIM WAS DROPPED WHEN THE STUDY WENT TO FULLY REMOTE DUE TO COVID
Description: The investigators will collect a single saliva sample at the end of the final night shift in the Baseline block and the Intervention block. The sample will be frozen and later assayed to assess cortisol level (in micrograms per deciliter, μg/dL). Higher cortisol levels will be indicative of greater stress.
Time Frame: Salivary Cortisol will be assessed immediately after the third night shift in the Intervention block and levels will be compared between groups.
Population: These data were not collected and therefore could not be analyzed. When the study had to go fully remote due to COVID, we dropped this Aim. This was reported in our NIH Progress Report in 2020.
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through each individual's study completion. This was from the start of data collection for an individual until the end of data collection for the individual, which was up to 4 weeks.
Description: No difference.
Arm/Group | Control (Group A) | 8-h Afternoon-Evening Sleep (Group B) | 8-h Free Sleep (Group C)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Group A) (N=10) | 8-h Afternoon-Evening Sleep (Group B) (N=10) | 8-h Free Sleep (Group C) (N=9)
acute shortness of breath (General disorders) | 1 (1) | 0 (0) | 0 (0) — The participant reported an incident of acute shortness of breath at the end of the baseline week. She underwent a stress echocardiogram which resulted in no adverse findings. She was cleared to return to work and completed the rest of the study.
motor vehicle accident (General disorders) | 0 (0) | 0 (0) | 1 (1) — Participant reported being rear-ended in a MVA on her way to work on the final night of the intervention week. Her airbags were deployed so she went to an ER to be evaluated. No injuries were sustained. She therefore did not work on that final night.

LIMITATIONS AND CAVEATS:
Enrollment in the study was hindered by the COVID-19 pandemic, and we had fewer participants than originally planned. We changed the study to be fully remote due to COVID and had to drop the salivary cortisol aim. Due to lower enrollment than planned, we could not address many of the secondary aims.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03813654/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03813654/ICF_001.pdf